CLINICAL TRIAL: NCT00050752
Title: Hereditary Leiomyomatosis Renal Cell Cancer (HLRCC): Identification of the Disease Gene, and Characterization of the Predisposition to Renal Cancer
Brief Title: Hereditary Leiomyomatosis Renal Cell Cancer - Study of the Genetic Cause and the Predisposition to Renal Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030066; 03-C-0066; NCT00055627 (obsolete NCT alias)
Record Dates: First submitted 2002-12-17; First posted 2002-12-18 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-07

CONDITIONS: Renal Tumor Histology; Cutaneous Leiomyoma; Kidney Cancer
Keywords: Renal Cancer; Hereditary Leiomyomatosis; Uterine Fibroid; Cutaneous Leiomyoma; Natural History
MeSH Terms: conditions — Kidney Neoplasms; Leiomyoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1 / Individuals: Individuals with known or suspected Hereditary Leiomyomatosis and Renal Cell Cancer Syndrome (HLRCC)
- 2 / Family Members: Family members (related by blood) of individuals who have or are suspected of having Hereditary Leiomyomatosis and Renal Cell Cancer Syndrome (HLRCC)
- 3 / Non-Biologic Family Members: Spouses enrolled primarily for linkage analysis (Spouses have been removed from the inclusion criteria for this study. This closed cohort is for spouses previously enrolled on study.)

SUMMARY:
This study will investigate what causes hereditary leiomyomatosis renal (kidney) cell cancer, or HLRCC, and how the disease is related to the development of kidney tumors. Leiomyomas are benign (non-cancerous) tumors arising from smooth muscle. HLRCC can cause various health problems. Some people develop red bumps on their skin that can be painful at times. Some women with HLRCC can develop leiomyomas of the uterus. In some families, people with HLRCC develop kidney tumors. This study will try to determine:

* What gene changes (mutations) cause HLRCC
* What kind of kidney tumors develop in HLRCC and how they grow
* What the chance is that a person with HLRCC will develop a kidney tumor

People with known or suspected HLRCC (and their family members of any age) may be eligible for this study. This includes people in families in which one or more members has skin leiomyoma and kidney cancer; skin leiomyoma and uterine leiomyoma; multiple skin leiomyomas; kidney cancer and uterine leiomyomas, or kidney cancer consistent with HLRCC, including, but not limited to, collecting duct or papillary, type II. Candidates will be screened with a physical examination, family history, and, for affected family members, a review of medical records, including pathology slides and computed tomography (CT) or magnetic resonance imaging (MRI) scans.

Participants will undergo tests and procedures that may include the following:

* Review of medical records, x-rays, and tissue slides
* Physical examination and family history
* Skin examination
* Gynecological examination for women
* Interviews with a cancer doctor, cancer nurses, kidney surgeon, and genetic counselor
* Blood tests for:

  1. Genetic research to identify the gene responsible for HLRCC
  2. Evaluation of liver, kidney, heart, pancreas, and thyroid function
  3. Complete blood count and clotting profile
  4. Pregnancy test for pre-menopausal women
  5. PSA test for prostate cancer in men over age 40
* CT or MRI scans (for participants 15 years of age and older only)
* Skin biopsy (surgical removal of a small sample of skin tissue)
* Cheek swab or mouth rinse to collect cells for genetic analysis
* Medical photographs of lesions
* Questionnaire

When the tests are completed, participants will discuss the results with a doctor and possibly a genetic nurse or genetic counselor. The genetic findings will not be revealed to participants because their meaning and implications may not yet be understood. Participants may be asked to return to NIH from every 3 months to every 3 years, depending on their condition, for follow-up examinations and tests.

DETAILED DESCRIPTION:
Background:

* Hereditary Leiomyomatosis and Renal Cell Cancer (HLRCC) is a rare autosomal dominantly inherited disorder which confers susceptibility to develop cutaneous and uterine leiomyomas and renal cell carcinoma.
* HLRCC is caused by mutations in the Krebs cycle enzyme, fumarate hydratase localized on chromosome 1q42.3-q43.

Objectives:

* Define the risk of developing renal cancer, cutaneous leiomyoma and uterine leiomyoma in this hereditary cancer syndrome
* Define the types and characteristics (including patterns of growth) of renal cancer associated with HLRCC
* Determine the incidence and characteristics of HLRCC-associated fumarate hydratase gene mutations
* Determine genotype/phenotype correlations
* Determine if other genes cause HLRCC

Eligibility:

* Individuals suspected or known to have phenotype or genotype suggestive of Hereditary Leiomyomatosis and Renal Cell Cancer Syndrome (HLRCC), such as individuals with:

  * Cutaneous leiomyoma and kidney cancer
  * Cutaneous leiomyoma and uterine leiomyoma
  * Multiple cutaneous leiomyoma
  * Kidney cancer and uterine leiomyomata
  * Renal tumor histology consistent with HLRCC including, but not limited to: Collecting Duct and/or Papillary, Type II
* A relative (related by blood) of an individual with a confirmed or suspected diagnosis of HLRCC

Design:

* These rare biological families will be recruited to genetically confirm diagnosis, determine size and location of renal tumors, size at presentation, growth rate and metastatic potential of renal tumors.
* Genetic testing will be offered to gain appreciation of the effect of mutations on the relative activity of various germline and somatic mutations.
* We will determine if there is a relationship between mutation and disease phenotype.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals suspected or known to have phenotype or genotype suggestive of Hereditary Leiomyomatosis and Renal Cell Cancer Syndrome (HLRCC), such as:

  * Cutaneous leiomyoma and kidney cancer; or
  * Cutaneous leiomyoma and uterine leiomyoma; or
  * Multiple cutaneous leiomyoma; or
  * Kidney cancer and uterine leiomyomata; or
  * Renal tumor histology consistent with HLRCC including, but not limited to: Collecting Duct and/or Papillary, Type II
* All participants and parents/guardians, for children younger than 18 years of age, must sign an informed consent document indicating their understanding of the investigational nature and the risks of this study before any protocol related studies are performed.
* Participants must be >= 2 years of age.
* A relative (related by blood) of an individual with a confirmed or suspected diagnosis of HLRCC.

EXCLUSION CRITERIA:

None

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: An individual (including patient) from a family in which one or more family member have: cutaneous leiomyoma and kidney cancer, cutaneous leiomyoma and uterine leiomyoma, multiple cutaneous leiomyoma, kidney cancer and uterine leiomyomata, renal tumor histology consistent with HLRCC including, but not limited to: Collecting Duct and/or Papillary, Type II.
Sampling Method: Non-Probability Sample
Enrollment: 1130 (Estimated)
Dates: Start 2003-02-24 (Actual)

PRIMARY OUTCOMES:
Determine the incidence and characteristics of HLRCC-associated fumarate hydratase gene mutations. | on-going
  Molecular genetic differences between normal and tumorigenic fumarate hydratase (fumerase) mutations.
Determine the clinical manifestations of HLRCC | on-going
  Collection of blood, urine and/or benign and malignant tissue.
Determine if other genes cause HLRCC. | on-going
  Molecular genetic differences between normal and tumorigenic cells.
Determine genotype/phenotype correlations. | on-going
  Detection and expression analysis of gene(s).
Define the types and characteristics (including patterns of growth) of renal cancer associated with HLRCC. | on-going
  Detection and expression analysis of gene(s).
Define the risk of developing renal cancer, cutaneous leiomyoma and uterine leiomyoma in this hereditary cancer syndrome. | on-going
  Collection of blood, urine and/or benign and malignant tissue.

CONTACTS AND LOCATIONS:
Overall Officials: W. Marston Linehan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Linehan WM, Lerman MI, Zbar B. Identification of the von Hippel-Lindau (VHL) gene. Its role in renal cancer. JAMA. 1995 Feb 15;273(7):564-70. No abstract available. PMID 7837390
- [Background] Latif F, Tory K, Gnarra J, Yao M, Duh FM, Orcutt ML, Stackhouse T, Kuzmin I, Modi W, Geil L, et al. Identification of the von Hippel-Lindau disease tumor suppressor gene. Science. 1993 May 28;260(5112):1317-20. doi: 10.1126/science.8493574.
- [Background] Zbar B, Tory K, Merino M, Schmidt L, Glenn G, Choyke P, Walther MM, Lerman M, Linehan WM. Hereditary papillary renal cell carcinoma. J Urol. 1994 Mar;151(3):561-6. doi: 10.1016/s0022-5347(17)35015-2. PMID 8308957
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2003-C-0066.html